CLINICAL TRIAL: NCT01450332
Title: A Single Arm, Prospective, Single Center, Study To Evaluate The Safety And Efficacy Of Tavor ACL Prosthesis In Patient With ACL Rupture
Brief Title: Safety and Efficacy of the Knee-T-nol Anterior Cruciate Ligament (ACL) Prosthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tavor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TACLPPS01 Rev 4
Record Dates: First submitted 2011-10-09; First posted 2011-10-12 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: ACL; arthroscopy; ligament; rupture; reconstruction; ACLR; accelerated rehabilitation program
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- study (Experimental)
  Interventions: Device: Knee-T-Nol

INTERVENTIONS:
Device: Knee-T-Nol — The ACL prosthesis is intended for the treatment of ruptured ACL. It will be used as an implant to replace the native, torn ACL. Implantation will be done using arthroscopy

SUMMARY:
The study is designed to evaluate the safety and efficacy of implanting the Tavor ACL prosthesis in patients with a ruptured ACL by improvement of healing kinetics as well as major adverse treatment events (AEs). it is designed to test the hypothesis that there is a difference in healing kinetics of ACL deficient knees treated by ACL reconstruction using autografts and those in which such procedure was performed with the Tavor prosthesis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is >= 18 years old
2. Patient has a ruptured ACL
3. Operated knee has full range of motion and no swelling
4. Patient understands the study requirements and the treatment procedures and rehabilitation and provides written Informed Consent before any study-specific tests or procedures are performed.
5. The patient commits to fully undergo the rehabilitation program and return for the scheduled post-operative follow-up visits at the clinic.

Exclusion Criteria:

1. Skeletal immaturity
2. Pregnancy
3. Patient with:

   * Uncontrolled systemic hypertension
   * Severe uncontrolled Diabetes Mellitus
   * Epiphyses That Have Not Yet Closed
   * Periarticular or Patella Fracture
   * History of Metabolic Bone Disease (e.g.., Osteoporosis, Rickets)
   * Crystal deposition disease, e.g., gout
   * Inflammatory joint disease, e.g., rheumatoid arthritis
   * Severe degenerative joint disease
   * Known neoplastic disease
   * HIV positive
   * Current steroid therapy in excess of prednisone 5 mg/day
   * Other severe, life-threatening systemic disease or any medical condition that interferes with their ability to participate in a rehabilitation program
4. The subject has participated in, or is planned to participate in, any investigational drug or device study within the past 30 days and for the duration of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Knee stability, as measured by a KT-1000 Arthrometer or Lachman test post procedure | post procedure
No treatment emergent SAEs, including Adverse Events of Interest (AEOI), 3 months post procedure. | 3 months post procedure

SECONDARY OUTCOMES:
Rehabilitation period, defined by Post procedure period [weeks] to successful rehabilitation phase | 3-6 months
  Rehabilitation period, defined by Post procedure period [weeks] to successful rehabilitation phase, as demonstrated by the ability of the patient to perform the following functional tests:
  * 70% of single leg 1 Rep Max on leg press vs. uninvolved
  * 10 single leg squats from 0-45° of flexion without loss of balance, muscle quivering, or varus/valgus moments (patella moving out of the sagittal plane)
  * 30 consecutive forward step-and-holds from the uninvolved to involved leg without loss of balance, muscle quivering, or varus/valgus moments (patella moving out of the sagittal plane)
Tegner Lysholm scores during the followup period | 12 months post op
  Short term Tegner Lysholm knee score >= 65, 3 months post procedure. Long term Knee stability, as measured by a KT-1000 Arthrometer or Lachman test at 12 months post procedure.
  Long term Tegner Lysholm knee score >= 84, 12 months post procedure. Procedure time, as compared to standard autograft procedure
Long term safety: no device related SAEs 12 months post procedure. | 12 months post op

CONTACTS AND LOCATIONS:
Overall Officials: Idan M Tobis, B.Sc., Study Director — Tavor Ltd.; Yoram Litwin, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shhare Zedek Medical Center, Jerusalem, Israel, Israel